CLINICAL TRIAL: NCT02454413
Title: ASSESSMENT OF THE IMPACT OF CLEANING METHODS AND OVERNIGHT DENTURE STORAGE ON BIOFILM FORMATION ON REMOVABLE ACRYLIC DENTURES.
Brief Title: Microbial Evaluation of Denture Cleaning and Overnight Storage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Joke Duyck, Professor, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2
Record Dates: First submitted 2013-01-15; First posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Denture Hygiene
Keywords: dentures hygiene; biofilm formation; oral health
MeSH Terms: interventions — Water; Soaps

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- brush + water (Sham Comparator): denture brushing with water and soap + overnight storage in water
  Interventions: Other: denture brushing with water and soap
- brush + cleansing tablet (Active Comparator): denture brushing with water and soap + overnight storage in water with a cleansing tablet
  Interventions: Other: denture brushing with water and soap; Other: cleansing tablet
- ultrasonic cleaning + water (Sham Comparator): ultrasonic denture cleaning + overnight storage in water
  Interventions: Other: ultrasonic denture cleaning
- ultrasonic cleaning + cleansing tablet (Active Comparator): ultrasonic denture cleaning + overnight storage in water with a cleansing tablet
  Interventions: Other: ultrasonic denture cleaning; Other: cleansing tablet

INTERVENTIONS:
Other: denture brushing with water and soap — denture brushing with water and soap
  Arms: brush + cleansing tablet; brush + water
Other: ultrasonic denture cleaning — ultrasonic denture cleaning
  Arms: ultrasonic cleaning + cleansing tablet; ultrasonic cleaning + water
Other: cleansing tablet — addition of a cleansing tablet to the water in which the dentures are stored overnight
  Arms: brush + cleansing tablet; ultrasonic cleaning + cleansing tablet

SUMMARY:
Clinical guidelines for denture care are available, but evidence for optimal nocturnal storage is missing. The investigators (Duyck J., Vandamme K., Teughels W.) therefore performed a study (submitted for publication) to evaluate the effect of different overnight storage protocols on denture biofilm formation and maturation. The results of this study showed that the use of cleansing tablets (Corega Tabs Anti-bacteria®, GlaxoSmithKline Consumer Healthcare SA, Genval, Belgium) for acrylic removable denture overnight storage reduces denture biofilm mass and pathogenicity compared to dry and water preservation. As no mechanical denture cleaning was performed in the aforementioned study, the aim of the proposed study is to evaluate the combined effect of mechanical cleaning and overnight storage condition on the microbial composition and Candida albicans colonization of denture biofilm formation. This information is required to develop a clinical guideline on acrylic denture cleaning and overnight storage aiming to reduce the risk posed by pathogenic microorganisms, particularly in bedridden and immunocompromised patients.

It is hypothetised that mechanical denture cleaning will decrease the impact of overnight denture storage condition on biofilm formation on acrylic removable dentures.

DETAILED DESCRIPTION:
Aim of the study

The presence of a biofilm - i.e. structured microbial communities that are attached to a surface and encased in an exopolymer matrix - on acrylic removable dentures has been associated with serious systemic conditions, especially in the dependent elderly [1]. Oral bacteria have been implicated in bacterial endocarditis [2], aspiration pneumonia [3, 4], chronic obstructive pulmonary disease [5, 6], amongst other diseases [1, 7]. Ample evidence is provided regarding the relationship between proper oral hygiene and overall systemic health.

Plaque on dentures is a complex aggregate containing more than 108 organisms per milligram, and involving more than 600 prokaryote species [8]. The different species collaborate to form a symbiotic biofilm. The biofilms in dentate patients have been studied extensively, but there have been few studies on the biofilm microbiota of complete acrylic dentures [10-18]. It appears that distinct biofilms, with associated pathogenic risks, are present in 'healthy' versus denture stomatitis affected participants [15, 16, 18]. Not only poor denture cleaning but also inappropriate habits, such as wearing dentures overnight have proved to be associated with the prevalence of Candida-associated stomatitis [19, 20]. Therefore, the overnight removal of the acrylic removable dentures is advised in clinical settings. Although evidence-based guidelines for denture care and maintenance are available [21], guidelines for nocturnal storage conditions of dentures are missing. The investigators therefore performed a study (submitted for publication) to evaluate the effect of different overnight storage protocols on denture biofilm formation and maturation. The results of this study showed that the use of cleansing tablets (Corega Tabs Anti-bacteria®, GlaxoSmithKline Consumer Healthcare SA, Genval, Belgium) for acrylic removable denture overnight storage reduces denture biofilm mass and pathogenicity compared to dry and water preservation.

As no mechanical denture cleaning was performed in the aforementioned study, the aim of the proposed study is to evaluate the combined effect of mechanical cleaning and overnight storage condition on the microbial composition and Candida albicans colonization of denture biofilm formation. This information is required to develop a clinical guideline on acrylic denture cleaning and overnight storage aiming to reduce the risk posed by pathogenic microorganisms, particularly in bedridden and immunocompromised patients.

Research questions

•What is the effect of mechanical cleaning on biofilm formation on removable acrylic dentures?

* Is ultrasonic cleaning more efficient compared to denture brushing with respect to prevention of biofilm formation on removable acrylic dentures?
* What is the effect of overnight storage in water with a cleansing tablet on biofilm formation on mechanically cleaned removable acrylic dentures?

Materials & Methods

* Participants -number: 30 -Inclusion criteria: Institutionalised frail elder Fully edentulous in lower and upper jaw Removable denture wearer in lower and upper jaw Good oral health

  -Exclusion criteria: Current or history of corticosteroid treatment within the 3 months prior to the study Current or history of antimicrobial treatment within the 3 months prior to the study Inability to provide informed consent Inability to comply with the study requirements
* Test conditions Denture cleaning method Denture overnight storage condition

  1Brushing with water and soap Immersion in water with a cleansing tablet 2Brushing with water and soap Immersion in water without a cleansing tablet (= neg control) 3Ultrasonic cleaning Immersion in water with a cleansing tablet 4Ultrasonic cleaning Immersion in water without a cleansing tablet
* This study was approved by the Institutional Ethics Committee (S54968, University Hospitals Leuven, Belgium) and registered in the Belgian Clinical Trials database (Identifier: B322201316863).
* Study design

  -Cross-over study with randomized sequence of the 4 test conditions This implies that all 4 test conditions will be executed within each of the 30 study participants.
  * The sequence of the test conditions for the individual participants will be randomized.
  * Double blind (both the participants as well as the investigators do not know the test conditions)
* All test conditions will be applied for 5 days. This means that all patients will undergo 4 test periods of 5 days.
* Each test period will be preceded by a wash-out period of 2 days in which the standard of care will be applied. This standard of care is denture cleaning through brushing with water and soap and overnight storage in water.
* All dentures will be decalcified using vinegar prior to the start of the study.
* At the start of the study, all dentures will be mechanically cleaned by means of denture brushing and additional ultrasonic cleaning. After mechanical cleaning, the dentures will also be desinfected using a 1% chlorhexidine digluconate gel (Corsodyl gel, GlaxoSmithKline Consumer Healthcare SA, Genval, Belgium).
* After mechanical denture cleaning and desinfection at the start of each test period, control samples (n=4) will be taken to evaluate the effectiveness of the cleaning and desinfection procedures.
* After each test period, test samples (n=4) will be taken
* The participants will be asked not to clean their dentures themselves. 2 care takers involved in the study will do the denture cleaning and will apply the appropriate overnight storage condition.
* Outcome measures:

Clinical health of the denture bearing mucosa Method: clinical evaluation Microbial analyses Method: qualitative and quantitative PCR analyses for 20 selected oral bacteria (Aa, Pg, Tf, Td, Pi, Fn, Pm, Pn, Cg, Cr, En, Ec, Cs, Cc, Sm, Sg, Sc, Ao, Av, Vp) and for Candida Albicans.

Biofilm sampling will be performed in a 5-mm diameter circular region of interest, situated bucco-distally to the lower second premolars (Figure 1). In order to standardize the position and dimensions of this region and to ensure optimal reproducibility of the microbial sampling, a custom-made mold of each lower prosthesis with placeholder rings will be made (Optosil®, Heraeus Kulzer GmbH, Hanau, Germany) (Figure 1). The placeholder rings will be placed in such a way that the transition between artificial teeth and gums is situated centrally. These molds will fabricated following denture disinfection at the start of the study, and will be re-used throughout the study because of the absence of dimensional changes over time when preserved properly (i.e. dry and in plastic bag). The molds and rings will be desinfected after each microbial sampling.

Denture plaque score Method: Denture plaque will be scored independently by 2 investigators using 4% erythrosine disclosing solution according to Augsburger and Elahi [22] (score range 0-4)

•Study protocol Time point Action Microbial sampling Day 0 (morning) calculus removal using vinegar mechanical denture cleaning ° Day 0-2 standard of carei Day 3 (morning) Mechanical denture cleaning° and desinfectionii control sample 1* Day 3-7 test period 1 Day 7 (evening) Mechanical denture cleaning° and desinfectionii test sample 1** Day 8-9 standard of carei (wash-out period) Day 10 (morning) Mechanical denture cleaning° and desinfectionii control sample 2* Day 10-14 test period 2 Day 14 (evening) Mechanical denture cleaning° and desinfectionii test sample 2** Day 15-16 standard of carei (wash-out period) Day 17 (morning) Mechanical denture cleaning° and desinfectionii control 3* Day 17-21 test period 3 Day 21 (evening) Mechanical denture cleaning° and desinfectionii test sample 3** Day 22-23 standard of carei (wash-out period) Day 24 (morning) Mechanical denture cleaning° and desinfectionii control 4* Day 24-28 test period 4 Day 28 (evening) Mechanical denture cleaning° and desinfectionii END OF THE STUDY test sample 4**

°mechanical denture cleaning: brushing with water and soap + additional ultrasonic cleaning i standard of care: denture brushing with water and soap and overnight storage in tab water iidesinfection with 1% chlorhexidine digluconate gel (Corsodyl gel, GlaxoSmithKline Consumer Healthcare SA, Genval, Belgium)

*control sampling: after mechanical cleaning and desinfection

**test sampling: before mechanical cleaning desinfection

ELIGIBILITY:
Inclusion Criteria:

* Institutionalised frail elder
* Fully edentulous in lower and upper jaw
* Removable denture wearer in lower and upper jaw
* Good oral health

Exclusion Criteria:

* Current or history of corticosteroid treatment within the 3 months prior to the study
* Current or history of antimicrobial treatment within the 3 months prior to the study
* Inability to provide informed consent
* Inability to comply with the study requirements

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Biofilm (quantity and quality) on the removable acrylic denture | sample taken at day 5 of the test period

SECONDARY OUTCOMES:
Oral health status | oral health control at day 5 of the test period

CONTACTS AND LOCATIONS:
Overall Officials: Joke JA Duyck, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

REFERENCES:
- [Background] Coulthwaite L, Verran J. Potential pathogenic aspects of denture plaque. Br J Biomed Sci. 2007;64(4):180-9. doi: 10.1080/09674845.2007.11732784. PMID 18236742
- [Background] Que YA, Moreillon P. Infective endocarditis. Nat Rev Cardiol. 2011 Jun;8(6):322-36. doi: 10.1038/nrcardio.2011.43. Epub 2011 Apr 12. PMID 21487430
- [Background] Raghavendran K, Mylotte JM, Scannapieco FA. Nursing home-associated pneumonia, hospital-acquired pneumonia and ventilator-associated pneumonia: the contribution of dental biofilms and periodontal inflammation. Periodontol 2000. 2007;44:164-77. doi: 10.1111/j.1600-0757.2006.00206.x. No abstract available. PMID 17474932
- [Background] El-Solh AA. Association between pneumonia and oral care in nursing home residents. Lung. 2011 Jun;189(3):173-80. doi: 10.1007/s00408-011-9297-0. Epub 2011 Apr 30. PMID 21533635
- [Background] Scannapieco FA. Pneumonia in nonambulatory patients. The role of oral bacteria and oral hygiene. J Am Dent Assoc. 2006 Oct;137 Suppl:21S-25S. doi: 10.14219/jada.archive.2006.0400. PMID 17012732
- [Background] Pace CC, McCullough GH. The association between oral microorgansims and aspiration pneumonia in the institutionalized elderly: review and recommendations. Dysphagia. 2010 Dec;25(4):307-22. doi: 10.1007/s00455-010-9298-9. Epub 2010 Sep 8. PMID 20824288
- [Background] Senpuku H, Sogame A, Inoshita E, Tsuha Y, Miyazaki H, Hanada N. Systemic diseases in association with microbial species in oral biofilm from elderly requiring care. Gerontology. 2003 Sep-Oct;49(5):301-9. doi: 10.1159/000071711. PMID 12920350
- [Background] Dewhirst FE, Chen T, Izard J, Paster BJ, Tanner AC, Yu WH, Lakshmanan A, Wade WG. The human oral microbiome. J Bacteriol. 2010 Oct;192(19):5002-17. doi: 10.1128/JB.00542-10. Epub 2010 Jul 23. PMID 20656903
- [Background] Mager DL, Ximenez-Fyvie LA, Haffajee AD, Socransky SS. Distribution of selected bacterial species on intraoral surfaces. J Clin Periodontol. 2003 Jul;30(7):644-54. doi: 10.1034/j.1600-051x.2003.00376.x. PMID 12834503
- [Background] Theilade E, Budtz-Jorgensen E, Theilade J. Predominant cultivable microflora of plaque on removable dentures in patients with healthy oral mucosa. Arch Oral Biol. 1983;28(8):675-80. doi: 10.1016/0003-9969(83)90101-2. PMID 6579900
- [Background] Moore TC, Smith DE, Kenny GE. Sanitization of dentures by several denture hygiene methods. J Prosthet Dent. 1984 Aug;52(2):158-63. doi: 10.1016/0022-3913(84)90087-8. PMID 6381698
- [Background] Koopmans AS, Kippuw N, de Graaff J. Bacterial involvement in denture-induced stomatitis. J Dent Res. 1988 Sep;67(9):1246-50. doi: 10.1177/00220345880670091901. PMID 3166009
- [Background] Chan EC, Iugovaz I, Siboo R, Bilyk M, Barolet R, Amsel R, Wooley C, Klitorinos A. Comparison of two popular methods for removal and killing of bacteria from dentures. J Can Dent Assoc. 1991 Dec;57(12):937-9. PMID 1760779
- [Background] Kononen E, Asikainen S, Alaluusua S, Kononen M, Summanen P, Kanervo A, Jousimies-Somer H. Are certain oral pathogens part of normal oral flora in denture-wearing edentulous subjects? Oral Microbiol Immunol. 1991 Apr;6(2):119-22. doi: 10.1111/j.1399-302x.1991.tb00463.x. PMID 1945487
- [Background] Campos MS, Marchini L, Bernardes LA, Paulino LC, Nobrega FG. Biofilm microbial communities of denture stomatitis. Oral Microbiol Immunol. 2008 Oct;23(5):419-24. doi: 10.1111/j.1399-302X.2008.00445.x. PMID 18793366
- [Background] Sachdeo A, Haffajee AD, Socransky SS. Biofilms in the edentulous oral cavity. J Prosthodont. 2008 Jul;17(5):348-56. doi: 10.1111/j.1532-849X.2008.00301.x. PMID 18355168
- [Background] Pereira-Cenci T, da Silva WJ, Cenci MS, Cury AA. Temporal changes of denture plaque microbiologic composition evaluated in situ. Int J Prosthodont. 2010 May-Jun;23(3):239-42. PMID 20552089
- [Background] Teles FR, Teles RP, Sachdeo A, Uzel NG, Song XQ, Torresyap G, Singh M, Papas A, Haffajee AD, Socransky SS. Comparison of microbial changes in early redeveloping biofilms on natural teeth and dentures. J Periodontol. 2012 Sep;83(9):1139-48. doi: 10.1902/jop.2012.110506. Epub 2012 Mar 23. PMID 22443543
- [Background] Compagnoni MA, Souza RF, Marra J, Pero AC, Barbosa DB. Relationship between Candida and nocturnal denture wear: quantitative study. J Oral Rehabil. 2007 Aug;34(8):600-5. doi: 10.1111/j.1365-2842.2007.01754.x. PMID 17650170
- [Background] Kulak-Ozkan Y, Kazazoglu E, Arikan A. Oral hygiene habits, denture cleanliness, presence of yeasts and stomatitis in elderly people. J Oral Rehabil. 2002 Mar;29(3):300-4. doi: 10.1046/j.1365-2842.2002.00816.x. PMID 11896849
- [Background] Felton D, Cooper L, Duqum I, Minsley G, Guckes A, Haug S, Meredith P, Solie C, Avery D, Deal Chandler N; American College of Prosthodontists. Evidence-based guidelines for the care and maintenance of complete dentures: a publication of the American College of Prosthodontists. J Prosthodont. 2011 Feb;20 Suppl 1:S1-S12. doi: 10.1111/j.1532-849X.2010.00683.x. PMID 21324026
- [Background] Augsburger RH, Elahi JM. Evaluation of seven proprietary denture cleansers. J Prosthet Dent. 1982 Apr;47(4):356-9. doi: 10.1016/s0022-3913(82)80079-6. No abstract available. PMID 6951034
- [Derived] Duyck J, Vandamme K, Krausch-Hofmann S, Boon L, De Keersmaecker K, Jalon E, Teughels W. Impact of Denture Cleaning Method and Overnight Storage Condition on Denture Biofilm Mass and Composition: A Cross-Over Randomized Clinical Trial. PLoS One. 2016 Jan 5;11(1):e0145837. doi: 10.1371/journal.pone.0145837. eCollection 2016. PMID 26730967